CLINICAL TRIAL: NCT02638194
Title: Adverse Health Effects of Mainstream and Secondhand Hookah Smoke in NYC Hookah Bars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-00370
Record Dates: First submitted 2015-12-11; First posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: COPD
Keywords: Chronic Obstructive Pulmonary Disease (COPD); smoking; secondhand smoke
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hookah Smoking Group (Active Comparator): 10 participants will smoke tobacco hookah for 2 hours
  Interventions: Other: Active smoking of Tobacco Hookah for 2 hours; Other: Visit a win bar
- Hookah Secondhand Smoke Group (Active Comparator): 10 individuals will be exposed to secondhand hookah tobacco smoke for 2 hours
  Interventions: Other: Exposure to tobacco hookah second hand smoke; Other: Visit a win bar

INTERVENTIONS:
Other: Active smoking of Tobacco Hookah for 2 hours
  Arms: Hookah Smoking Group
Other: Exposure to tobacco hookah second hand smoke
  Arms: Hookah Secondhand Smoke Group
Other: Visit a win bar — Participants will visit a wine bar for food and/or drinks

SUMMARY:
The primary purpose of this study is to examine the health effects of mainstream and secondhand hookah (i.e. water pipe) smoke on pulmonary and cardiovascular functions as well as serum levels of inflammatory biomarkers. Investigators would like to demonstrate that inhalation of both mainstream and secondhand smoke generated by hookah produces adverse pulmonary and cardiovascular effects and alterations in serum levels of inflammatory biomarkers.

DETAILED DESCRIPTION:
A total of 20 participants are going to be enrolled in this study; 10 participants smoke hookah and 10 participants are exposed to second hand hookah smoke for 2 hours in NYC hookah bars. Subjects in the control group will also be paired as they were for the hookah bar visit but will visit a control location, where they will be asked to consume a similar amount of food and drink at a wine bar. Pulmonary function, cardiovascular changes, and blood and urine markers of inflammatory mediators before, immediately after and 24 hours after the participants' visits to hookah bars and wine bars will be examined. Air quality monitoring will also be performed at the hookah bar and at the control location. Physiological changes will be assessed by measuring pulmonary function, blood pressure, heart rate, and blood oxygenation status. To determine the extent of tobacco exposure and associated inflammatory changes from secondhand hookah smoke, investigators will measure blood inflammatory biomarkers, oxidative stress, gene expression, tobacco-related carcinogenic metabolites, and exhaled carbon dioxide levels.

ELIGIBILITY:
Inclusion Criteria:

* Competent adult English speaking subjects
* Have used hookah in the past

Exclusion Criteria:

* Age <21
* Pregnancy
* Current cigarette smokers
* Has pulmonary disease, such as asthma or Chronic Obstructive Pulmonary Disease (COPD)
* Subjects are unable to give voluntary informed consent because they are non English speaking, are unable to read or write, or any other impediments that prohibits giving written informed consent
* Recent nasal surgery (within 6 months)
* History of bleeding or other blood related disorder.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes in exhaled carbon dioxide measured by pulmonary function measure using a portable spirometer | subsequently after 2 hours of hookah smoking or smoke exposure and 24 hours after participants' visit hookah and wine bars.
Changes in Heart Rate measured by a portable monitor worn during encounters | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in blood oxygenation levels measured by a pulse oximeter | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of tobacco-related carcinogenic metabolite cotinine in saliva samples | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of blood inflammatory marker endothelin | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of blood inflammatory marker IL-10 | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of blood inflammatory marker IL-8 | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of blood inflammatory marker IL-6 | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of blood inflammatory marker CRP | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of blood inflammatory marker IL-1a | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of blood inflammatory marker IFN-g | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of blood inflammatory marker TNF-a | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of blood inflammatory marker GM-CSF | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of blood inflammatory marker E-selectin | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of blood inflammatory marker thrombomodulin | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.
Changes in measure of blood inflammatory marker vWF | subsequently after 2 hours of hookah smoking and 24 hours after participants' visit hookah and wine bars.

SECONDARY OUTCOMES:
Changes in Air Quality measured by an aethelometer | 2 hours spent at hookah bar

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weitzman, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No